CLINICAL TRIAL: NCT00613574
Title: RUSSE / Russian Spiriva® Safety & Efficacy Study
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Other Study IDs: 205.396
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: tiotropium-bromide — Spiriva® inhaled capsule 18 mcg once daily administered via HandiHaler® on the top of usual care

SUMMARY:
At the moment, there is hardly any structured safety and efficacy data collection on Tiotropium in Russia. Therefore, the objective of this observational study is to collect and evaluate data on bronchodilator efficacy and safety of Spiriva® (18 µg tiotropium inhalation capsules) delivered by HandiHaler®, in a national sample of Russian patients with varying severities of chronic obstructive pulmonary disease (COPD) in a real life setting over the 8 weeks.

DETAILED DESCRIPTION:
The objective of this observational study is to collect and evaluate data on bronchodilator efficacy and safety of Spiriva® (18 µg tiotropium inhalation capsules) delivered by HandiHaler®, in national sample of Russian patients with varying severities of chronic obstructive pulmonary disease (COPD) in the real life setting over the 8 weeks.

Study Hypothesis:

Primary interest is given to observe change from baseline in post-dose FEV1 after 8 weeks.

Comparison(s):

The objective of this observational study is to collect and evaluate data on bronchodilator efficacy and safety of Spiriva® (18 mcg tiotropium inhalation capsules) delivered by HandiHaler®, in national sample of Russian patients with varying severities of chronic obstructive pulmonary disease (COPD) in a real life setting over the 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. 40 years and older male and female ambulatory outpatients being seen in a participating physicians office for routine care
2. Patients not previously treated with the Tiotropium
3. Patients with clinical diagnosis of all stages of Chronic Obstructive Pulmonary Disease according to the current National Guidelines / 2004
4. Current smokers or ex-smokers with a smoking history of >=10 pack years

Exclusion Criteria:

1. Uncooperative patients as judged by the physician,
2. Patients that have any condition which, according to the participating physicians opinion, might decrease the chance of obtaining satisfactory data to achieve the objectives of the observation,
3. Patients with history of known preexisting or concomitant non-obstructive lung disease (e.g., sarcoidosis, tuberculosis, lung cancer),
4. Patients currently enrolled in another clinical trial which requires a change in medication for their respiratory problems,
5. Patients with any conditions listed in special precautions, drug interactions, and contraindication of Spiriva®'s Russian package insert, such as:
6. Patients with known narrow-angle glaucoma,
7. Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction,
8. Patient with known moderate to severe renal impairment (creatinine clearance less than 50 ml/min),
9. Patients with a history of hypersensitivity to atropine or its derivatives, e.g. ipratropium or oxitropium or to any component of this product,
10. Pregnant or nursing women.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physicians
Sampling Method: Probability Sample
Enrollment: 407 (Actual)
Dates: Study Completion 2007-10

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — BI Pharma Ges mbH Wien
Locations (33):
- Russia (33):
  - Boehringer Ingelheim Investigational Site, Barnaul
  - Boehringer Ingelheim Investigational Site, Chelyabinsk
  - Boehringer Ingelheim Investigational Site, Irkutsk
  - Boehringer Ingelheim Investigational Site, Kazan'
  - Boehringer Ingelheim Investigational Site, Kemerovo
  - Boehringer Ingelheim Investigational Site, Khabarovsk
  - Boehringer Ingelheim Investigational Site, Krasnodar
  - Boehringer Ingelheim Investigational Site, Krasnodar Region
  - Boehringer Ingelheim Investigational Site, Krasnoyarsk
  - Boehringer Ingelheim Investigational Site, Kursk
  - Boehringer Ingelheim Investigational Site, Mezjdurechensk
  - Boehringer Ingelheim Investigational Site, Moscow
  - Boehringer Ingelheim Investigational Site, Moscow Region
  - Boehringer Ingelheim Investigational Site, Nizhny Novgorod
  - Boehringer Ingelheim Investigational Site, North Ossetia
  - Boehringer Ingelheim Investigational Site, Novosibirsk
  - Boehringer Ingelheim Investigational Site, Omsk
  - Boehringer Ingelheim Investigational Site, Perm
  - Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - Boehringer Ingelheim Investigational Site, Ryazan
  - Boehringer Ingelheim Investigational Site, S-Petersburg
  - Boehringer Ingelheim Investigational Site, Samara
  - Boehringer Ingelheim Investigational Site, Saratov
  - Boehringer Ingelheim Investigational Site, Stavropol
  - Boehringer Ingelheim Investigational Site, Stavropol Region, North Ossetia
  - Boehringer Ingelheim Investigational Site, Tomsk
  - Boehringer Ingelheim Investigational Site, Tyumen
  - Boehringer Ingelheim Investigational Site, Ufa
  - Boehringer Ingelheim Investigational Site, Vladivostok
  - Boehringer Ingelheim Investigational Site, Volgograd
  - Boehringer Ingelheim Investigational Site, Voroneg
  - Boehringer Ingelheim Investigational Site, Yaroslavl
  - Boehringer Ingelheim Investigational Site, Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Groups:
- Spiriva® (Tiotropium Bromide): Tiotropium bromide 18µg inhalation capsules once-daily
Period: Overall Study
Arm/Group | Spiriva® (Tiotropium Bromide)
Started | 407
Completed | 401
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 2
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Spiriva® (Tiotropium Bromide)
Number analyzed (Participants) | 407
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 339

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Post-dose Forced Expiratory Volume in 1 Second After 8 Weeks
Description: Forced expiratory volume in 1 second (FEV1) post-dose response at the end of the observation (Visit 3/week 8) versus (vs.) baseline (Visit 1/week 0)
Time Frame: baseline and final visit (8 weeks)
Population: Full Analysis Set (Intent-to-Treat population)
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Spiriva® (Tiotropium Bromide)
Number analyzed (Participants) | 401
liters | 0.29 (0.43)

2. Secondary Outcome: Change From Baseline for Forced Vital Capacity After 8 Weeks
Description: Forced vital capacity (FVC) post-dose response at end of the observation (Visit 3/week 8 ) vs. baseline (Visit 1/week 0)
Time Frame: baseline and final visit (8 weeks)
Population: Full Analysis Set (Intent-to-Treat population)
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Spiriva® (Tiotropium Bromide)
Number analyzed (Participants) | 401
liters | 0.31 (0.54)

3. Secondary Outcome: Change From Baseline for Inspiratory Capacity (*Only Selected Sites) After 8 Weeks
Description: Inspiratory capacity (IC) post-dose response at end of the observation (Visit 3/week 8) vs. baseline (Visit 1/week 0) at selected sites
Time Frame: Visit 1 to Visit 3 (baseline and 8 weeks)
Population: Full Analysis Set (Intent-to-Treat population) and only patients from selected sites
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Spiriva® (Tiotropium Bromide)
Number analyzed (Participants) | 245
liters | 0.18 (0.56)

4. Secondary Outcome: Patients Global Clinical Assessment of Efficacy at Final Visit by Severity, Full Analysis Set (FAS)
Description: Patient Global Assessment of Spiriva® efficacy with a 4-point scale (1=excellent efficacy&tolerability, 4=poor) at end of the observation (Visit 3/week 8).
Time Frame: final visit (8 weeks)
Population: Full Analysis Set (Intent-to-Treat population)
Measure: Number; unit: participants
Arm/Group | Spiriva® (Tiotropium Bromide)
Number analyzed (Participants) | 401
participants
  Excellent | 141
  Good | 198
  Satisfactory | 60
  Poor | 2

5. Secondary Outcome: Patients Global Clinical Assessment of Tolerability at Final Visit by Severity, FAS
Description: Patient Global Assessment of Spiriva® tolerability with a 4-point scale (1=excellent efficacy&tolerability, 4=poor) at end of the observation (Visit 3/week 8).
Time Frame: final visit (8 weeks)
Population: Full Analysis Set (Intent-to-Treat population)
Measure: Number; unit: participants
Arm/Group | Spiriva® (Tiotropium Bromide)
Number analyzed (Participants) | 401
participants
  Excellent | 246
  Good | 139
  Satisfactory | 16
  Poor | 0

6. Secondary Outcome: Physicians Global Clinical Assessment of Effect at Final Visit by Severity, FAS
Description: Physician Global Assessment of Spiriva® efficacy with a 4-point scale (1=excellent efficacy&tolerability, 4=poor) at end of the observation (Visit 3/week 8).
Time Frame: final visit (8 weeks)
Population: Full Analysis Set (Intent-to-Treat population)
Measure: Number; unit: participants
Arm/Group | Spiriva® (Tiotropium Bromide)
Number analyzed (Participants) | 401
participants
  Excellent | 159
  Good | 195
  Satisfactory | 45
  Poor | 2

7. Secondary Outcome: Physicians Global Clinical Assessment of Tolerability at Final Visit by Severity, FAS
Description: Physician Global Assessment of Spiriva® tolerability with a 4-point scale (1=excellent efficacy&tolerability, 4=poor) at end of the observation (Visit 3/week 8).
Time Frame: final visit (8 weeks)
Population: Full Analysis Set (Intent-to-Treat population)
Measure: Number; unit: participants
Arm/Group | Spiriva® (Tiotropium Bromide)
Number analyzed (Participants) | 401
participants
  Excellent | 246
  Good | 144
  Satisfactory | 11
  Poor | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Spiriva® (Tiotropium Bromide)
Serious Adverse Events (participants affected / at risk) | 2/407
Other Adverse Events (participants affected / at risk) | 0/407
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spiriva® (Tiotropium Bromide) (N=407)
Blastoma of Larynx (Respiratory, thoracic and mediastinal disorders) | 1
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.